CLINICAL TRIAL: NCT05508984
Title: Observational Study of Clinical Outcomes and Patient Satisfaction With Use of the Amma System
Brief Title: Clinical Outcomes and Patient Satisfaction With Use of the Amma System
Status: Active, not recruiting | Type: Observational
Sponsor: Providence Health & Services (Other)
Collaborators: Cooler Heads (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2022000438
Record Dates: First submitted 2022-08-11; First posted 2022-08-19 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
Keywords: Amma, Cooler Heads
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Single Arm: Anywhere from 14 to 0 days prior to treatment, enrolled subjects will complete the following questionnaires, and their hair will be photographed by research staff.
  Once enrolled, subjects will be provided the Amma device by the clinic on days of chemotherapy treatment, and upon completion of treatment it will be returned to the clinic for safekeeping. Upon completion of chemotherapy, anywhere from 3-6 weeks following treatment, subjects will repeat the questionnaires and their hair will be photographed again.
  Subjects will then complete their enrollment in the study.
  Interventions: Device: Amma Cooling Caps

INTERVENTIONS:
Device: Amma Cooling Caps — Once enrolled, subjects will be provided the Amma device by the clinic on days of chemotherapy treatment, and upon completion of treatment it will be returned to the clinic for safekeeping. Upon completion of chemotherapy, anywhere from 3-6 weeks following treatment, subjects will repeat the questionnaires and their hair will be photographed again.
  The overall duration of the study for subjects will be anywhere from 4 months to 8 months, depending on the duration of their chemotherapy regimen.

SUMMARY:
The primary goal is to conduct a pilot evaluation of the Amma device, to determine whether it is feasible to offer as an option for patients within oncology suites within the PH&S system.

DETAILED DESCRIPTION:
A novel cold capping device, named Amma™, is now commercially available for use and FDA approved. The Amma system has the potential to be as effective as the Penguin Cold Cap system, but with key innovations that make it more efficient and feasible in the clinic. Innovations include:

* Portable and battery powered unit, not requiring dry ice
* Form-fitting scalp cap that eliminates the need for frequent cap exchanges The Amma system has not been evaluated for efficacy, and no clinical trials are published.

Because of the ease of use and the self-directed administration of the Amma scalp cooling device, we wish to explore this as an option for patients treated within the PH&S system. To do this, we propose an observational study that evaluates clinical outcomes and patient-reported satisfaction amongst a cohort of patients who undergo self-directed scalp cooling using the Amma system.

ELIGIBILITY:
Inclusion Criteria:

- Women with stage I-III breast cancer are eligible to participate if:

* They consent to conduct baseline (week 0) and follow-up (week 4 post-chemo) surveys/interviews
* They consent to be photographed at baseline (week 0) and follow-up (week 4 post-chemo), to document hair retention outcomes
* Curative-intent chemotherapy is planned with a taxane-based, anthracycline-sparing chemotherapy regimen (which includes but may not be limited to: TC x 4, T x 12, TCHP x6)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with stage I-III breast cancer are eligible to participate.
Study Population: Women with stage I-III breast cancer are eligible to participate if they have a curative-intent chemotherapy regimen.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
AMMA Feasibility Within PH&S System | End of Treatment (4 to 8 months, depending on duration of their chemotherapy regimen)
  The primary goal is to conduct a pilot evaluation of the Amma device, to determine whether it is feasible to offer as an option for patients with early-stage breast cancer within oncology suites within the PH&S system. Patient satisfaction will be assessed using pre and post treatment questionnaires related to the Amma system and an exit interview.

SECONDARY OUTCOMES:
Patient Reported Outcome Utilizing Dean's Score | End of Treatment (4 to 8 months, depending on duration of their chemotherapy regimen)
  Patient satisfaction will be assessed via alopecia assessment utilizing Deans Scale collected at baseline and at end of treatment.
Patient Reported Outcome Utilizing Body Image Scale | End of Treatment (4 to 8 months, depending on duration of their chemotherapy regimen)
  Patient satisfaction will be assessed utilizing the Body Image Scale (BIS) questionnaire.
Patient Satisfaction Utilizing the Was It Worth It Questionnaire | End of Treatment (4 to 8 months, depending on duration of their chemotherapy regimen)
  Patient satisfaction will be assessed utilizing the Was It Worth It (WIWI) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: David Page, MD, Principal Investigator — Providence Health & Services
Locations (3):
- United States (3):
  - Providence Cancer Institute - Newberg Clinic, Newberg, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Oncology and Hematology Care - Westside, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No